CLINICAL TRIAL: NCT06594510
Title: AYANDRA Study: Addressing Youth and Adolescent Needs in Development, Research, and Advocacy
Brief Title: the Challenges of Young Adults With Cancer
Acronym: AYANDRA
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID 7061
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: AYA Cancer Patients; AYA Cancer Survivors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to describe unmet needs of Adolescent & Young Adults (AYA) with gastrointestinal and breast cancers in relation to: a) quality of life, b) education, c) finances and Insurance, and d) childbearing and parenting in Europe

DETAILED DESCRIPTION:
An electronic online questionnaire was developed addressing four main areas: a) quality of life, b) education, c) finances and Insurance, and d) childbearing and parenting. In brief, the first part of the questionnaire will aim to examine the demographic characteristics of the participants, such as their nationality, gender, age at diagnosis, actual age, and level of education, followed by their diagnosis or condition. No clinical data will be collected other than these features. Then, each domain will include 10 questions (multiple choice questions, ranking questions and 7-point Likert scale questions) and investigate the unmet needs in AYA with gastrointestinal and breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old at survey participation, as long as aged 13-39 years old at diagnois;
* Gastrointestinal cancer (colorectal, gastric, pancreatic) or breast cancer.

Exclusion Criteria:

* Age: 18 years old at survey participation;
* Patients 13 - 39 years old at diagnosis;
* Hematologic malignancies or different cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adolescent and Young Adults with gastrointestinal and breast cancers aged 13-39 -years old at diagnosis.
Sampling Method: Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
AYA Quality of life (QoL) | From answering to the end of the survey after 15 minutes
  Assessed by the EQ-5D-5L index and the descriptive statistic of the unmet needs in relation to the 4 domains of investigation, : a) quality of life, b) education, c) finances and Insurance, and d) childbearing and parenting
AYA Education | From answering to the end of the survey after 15 minutes
  Assessed by the descriptive statistic of the unmet needs obtained from the survey in relation to the 4 domains of investigation.
AYA Finances and Insurance | From answering to the end of the survey after 15 minutes
  Assessed by the descriptive statistic of the unmet needs obtained from the survey in relation to the 4 domains of investigation.
AYA Childbearing and Parenting | From answering to the end of the survey after 15 minutes
  Assessed by the descriptive statistic of the unmet needs obtained from the survey in relation to the 4 domains of investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Lorenzon, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Chirurgia Generale 1, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nichols HB, Baggett CD, Engel SM, Getahun D, Anderson C, Cannizzaro NT, Green L, Gupta P, Laurent CA, Lin PC, Meernik C, Moy LM, Wantman E, Xu L, Kwan ML, Mersereau JE, Chao CR, Kushi LH. The Adolescent and Young Adult (AYA) Horizon Study: An AYA Cancer Survivorship Cohort. Cancer Epidemiol Biomarkers Prev. 2021 May;30(5):857-866. doi: 10.1158/1055-9965.EPI-20-1315. Epub 2021 Feb 22. PMID 33619021
- [Result] Stoneham SJ. AYA survivorship: The next challenge. Cancer. 2020 May 15;126(10):2116-2119. doi: 10.1002/cncr.32774. Epub 2020 Mar 4. No abstract available. PMID 32129904
- [Result] Ferrari A, Stark D, Peccatori FA, Fern L, Laurence V, Gaspar N, Bozovic-Spasojevic I, Smith O, De Munter J, Derwich K, Hjorth L, van der Graaf WTA, Soanes L, Jezdic S, Blondeel A, Bielack S, Douillard JY, Mountzios G, Saloustros E. Adolescents and young adults (AYA) with cancer: a position paper from the AYA Working Group of the European Society for Medical Oncology (ESMO) and the European Society for Paediatric Oncology (SIOPE). ESMO Open. 2021 Apr;6(2):100096. doi: 10.1016/j.esmoop.2021.100096. PMID 33926710
- [Result] Miller KD, Fidler-Benaoudia M, Keegan TH, Hipp HS, Jemal A, Siegel RL. Cancer statistics for adolescents and young adults, 2020. CA Cancer J Clin. 2020 Nov;70(6):443-459. doi: 10.3322/caac.21637. Epub 2020 Sep 17. PMID 32940362
- [Result] Pilozzi E, Lorenzon L, Lo Baido S, Ferri M, Duranti E, Fochetti F, Mercantini P, Ramacciato G, Balducci G, Ruco L. Left-sided early onset colorectal carcinomas: A sporadic neoplasm with aggressive behavior. Am J Surg. 2017 Sep;214(3):421-427. doi: 10.1016/j.amjsurg.2017.01.035. Epub 2017 Jan 31. PMID 28173936